CLINICAL TRIAL: NCT04895085
Title: ReSET Aim 1a: Restarting Safe Education and Testing for Children With Medical Complexity - Feasibility of In-home Cohort SARS-CoV-2 Testing Strategies, and Associations With CMC Parent Perceptions About In-person School Attendance
Brief Title: ReSET Aim 1a: Restarting Safe Education and Testing for Children With Medical Complexity - Feasibility of In-home Cohort COVID-19 Testing Strategies, and Associations With CMC Parent Perceptions About In-person School Attendance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-0462; 1OT2HD107558-01 (NIH); A536771 (Other: UW, Madison); SMPH/PEDIATRICS (Other: UW, Madison); Protocol Version 04/12/21 (Other: UW Madison); 2022-0594 (Other: UW Madison)
Record Dates: First submitted 2021-05-14; First posted 2021-05-20 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: COVID-19; Children With Medical Complexity (CMC)
Keywords: Caregiver; in-person school attendance; In-home COVID testing
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is a single site study taking place over 24 months and involving (50) caregivers and their children with medical complexity. Additionally, (20) of these caregivers will be invited to participate in an hour-long, virtual contextual inquiry session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Caregiver of Children with medical complexity (CMC) (Experimental)
  Interventions: Diagnostic Test: BinaxNOW Rapid Antigen System

INTERVENTIONS:
Diagnostic Test: BinaxNOW Rapid Antigen System — BinaxNOW Rapid Antigen System (Abbott) is a point-of-care, lateral flow immunoassay intended for the qualitative detection of nucleocapsid protein antigen from SARS-CoV-2 in direct anterior nasal (nares) swabs. Internal controls are built into the testing system and results are available in 15 minutes.
  The use of the BinaxNOW system is authorized under the Food and Drug Administration's Emergency Use Authorization. The test is allowed for over-the-counter, non-prescription use with or without symptoms. The test may be used with children two years and older with the help of sample collection by an adult, and the test may be self-administered by anyone aged 15 years or more.

SUMMARY:
The purpose of this research study is to learn about the factors parents consider when deciding whether their child will go to school in-person or attend from home. Investigators are also interested in learning whether access to in-home COVID testing is of value to parents and also whether it affects decision-making about returning to school.

This study is being done at UW-Madison in partnership between the Department of Pediatrics and the Department of Industrial and Systems Engineering. A total of 50 caregivers (plus their children with medical complexity) will participate in this study. Additionally, 20 caregivers involved in the study may also be invited to participate in a one-hour, virtual visit in which the caregiver demonstrates and discusses how they perform in-home COVID testing with their child.

The results of the study may help researchers advance their understanding of in-home testing strategies for children with medical complexity.

DETAILED DESCRIPTION:
During the first three months of the study, caregivers will be asked to perform the BinaxNOW Rapid Antigen test on their child twice-weekly. After the first three months of the study, the testing schedule will depend on the statewide (WI) community spread rate. If the rate of spread is above the threshold for higher risk of transmission in schools (defined by the CDC as ≥ 25 new cases per 100,000 population in past 7 days) caregivers will be asked to continue twice-weekly surveillance. If it is below the threshold, caregivers will be offered the option to continue twice-weekly testing or switch to symptomatic-only testing. The study staff will notify caregivers of changes in testing frequency during their weekly communication. Caregivers will be asked to document their testing activities, results, and any possible COVID-19 symptoms on a Parent Testing Log.

If testing produces a negative result, the caregiver will be instructed to document the test result on their testing log. While false negative tests are possible with asymptomatic individuals, there will be no change in standard mitigation measures based on the test results (mandatory masks in school, social distancing, hand hygiene, etc.).

If testing produces a positive result from an asymptomatic individual, the caregiver will be instructed to contact the study team immediately and then obtain a PCR (polymerase chain reaction) test within 48 hours. The study staff will assist the caregiver in making arrangements for this test. In the case of positive tests, children will be restricted from school activities per public health guidelines until the results of the PCR testing are known. If the PCR test returns as a negative result and the child is attending school in-person, they will be allowed to return to school the next day (or if symptomatic, once symptoms resolve). If the PCR returns as positive, the caregiver will be instructed to keep the child at home per public health guidelines. To support families and ensure these steps occur, the study staff will call families daily following positive tests.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, the caregiver/child must meet the following criteria:

* The caregiver is willing to comply with all study procedures and expects to be available for the duration of the study.
* The caregiver is at least 18 years of age.
* The caregiver is proficient in English.
* The caregiver is self-identified as the primary caregiver (parent, foster parent, legal guardian) of a CMC who is aged 5-16 years at the start of the study and who is enrolled in the Pediatric Complex Care Program (PCCP) at the University of WI-Madison.
* The caregiver is currently providing care on an ongoing basis to their CMC. The child may not be housed in a skilled nursing facility, an acute care or transitional facility, a rehabilitative hospital, a medical group home or in a foster home (unless the primary caregiver for the study is the foster parent).
* The caregiver has access to a web-enabled device (phone, tablet, or computer).
* Caregiver and child are residents of Wisconsin.
* The child attended in-person school pre-pandemic. (Child can currently be attending school in-person, remotely or a hybrid combination).
* The caregiver provides a written informed consent form.

Exclusion Criteria:

* Failure to meet all inclusion criteria.
* The child is hospitalized at the time of enrollment (visit may be rescheduled)
* Children not currently enrolled in public or private school and whose caregiver has no plan to enroll them in the Fall of 2021 (e.g., children currently homeschooling with plans to homeschool in the Fall of 2021 are ineligible).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Coller, MD, MPH, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol enrollment, started, and completed values reflect caregiver/child dyads. All dyads assigned to the intervention had one caregiver to one child (n = 51 caregivers, n = 51 children). All participants were assigned to the intervention group.
Period: Overall Study
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Started | 51 (Caregiver/child dyads where caregiver n = 51 and child n = 51.)
Completed | 48 (Caregiver/child dyads where caregiver n = 48 and child n = 48.)
Not Completed | 3
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — No longer eligible: Moved from area | 1

BASELINE CHARACTERISTICS:
Population: All data was collected from caregivers.
Groups:
- Child With Medical Complexity: BinaxNOW Rapid Antigen System: BinaxNOW Rapid Antigen System (Abbott) is a point-of-care, lateral flow immunoassay intended for the qualitative detection of nucleocapsid protein antigen from SARS-CoV-2 in direct anterior nasal (nares) swabs. Internal controls are built into the testing system and results are available in 15 minutes.
  The use of the BinaxNOW system is authorized under the Food and Drug Administration's Emergency Use Authorization. The test is allowed for over-the-counter, non-prescription use with or without symptoms. The test may be used with children two years and older with the help of sample collection by an adult, and the test may be self-administered by anyone aged 15 years or more.
- Total: Total of all reporting groups
Arm/Group | Caregiver of Children With Medical Complexity (CMC) | Child With Medical Complexity | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 51 | 51
  Between 18 and 65 years | 51 | 0 | 51
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 39 [35 to 41] | 9 [6 to 12] | NA [NA to NA] — Two separate groups. Not applicable to analyze together.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 20 | 68
  Male | 3 | 31 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 46 | 44 | 90
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 46 | 42 | 88
  More than one race | 0 | 4 | 4
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51 | 51 | 102

OUTCOME MEASURES:

1. Primary Outcome: Change in Protocol Uptake: Number of Participants Consented Compared to Number of Participants Approached
Description: Feasibility of home based COVID-19 testing will be evaluated by protocol uptake. Data will be retrieved from the study log.
Time Frame: Study duration (up to 21 months)
Population: The number of participants analyzed must reflect the number of participants approached in addition to those consented.
Measure: Number; unit: Caregiver/child dyads
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 84
Caregiver/child dyads
  Number approached, consented | 51
  Number approached, not consented | 33

2. Primary Outcome: Change in Mean Number of Weekly in Home COVID-19 Tests
Description: Feasibility of home based COVID-19 testing will be evaluated by the mean number of weekly in home COVID-19 tests run by parents/caregivers. Data will be collected by survey.
Time Frame: Every week up to 21 months
Measure: Mean (Standard Deviation); unit: BinaxNow Antigen COVID-19 Tests per week
Units Other Than Participants: BinaxNOW Rapid Antigen COVID-19 Tests
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Number analyzed (BinaxNOW Rapid Antigen COVID-19 Tests) | 3254
BinaxNow Antigen COVID-19 Tests per week | 1.8 (0.3)

3. Primary Outcome: Change in COVID Test Rate at Home: Number of Total Tests Completed as Compared to Number of Tests Expected
Description: Data will be collected by survey.
  * Tests expected: Various scenarios factor into the tests expected value. Caregivers were expected to test their child twice a week every week for the first three months. After that time, caregivers could opt-in to surveillance testing (expected testing twice a week every week) or proceed with symptomatic-only testing (no "expected" tests for caregivers). Additionally, caregivers were not expected to test for 90 days after their child tested positive.
  * Tests completed: Caregivers were allowed to test more often than twice a week if appropriate (e.g., exposure to COVID-19). All symptomatic-only tests were not considered expected tests. These factors allowed the number of tests completed to exceed the number of tests expected.
Time Frame: Study duration (up to 21 months)
Measure: Number; unit: BinaxNOW Rapid Antigen COVID-19 Tests
Units Other Than Participants: BinaxNOW Rapid Antigen COVID-19 Tests
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Number analyzed (BinaxNOW Rapid Antigen COVID-19 Tests) | 3254
BinaxNOW Rapid Antigen COVID-19 Tests
  Number of tests completed | 3254
  Number of tests expected | 2572

4. Primary Outcome: Change in Symptomatic Test Rate: Number of Symptomatic Tests Completed
Description: Data will be collected from parents via survey.
Time Frame: Study duration (up to 21 months)
Measure: Number; unit: Symptomatic BinaxNow Rapid Antigen Tests
Units Other Than Participants: BinaxNOW Rapid Antigen COVID-19 Tests
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Number analyzed (BinaxNOW Rapid Antigen COVID-19 Tests) | 3254
Symptomatic BinaxNow Rapid Antigen Tests | 729

5. Primary Outcome: Change in Positive Rate: Number of Positive COVID-19 Tests Compared to Total Number of Tests Performed
Description: Data will be collected from parents via survey.
Time Frame: Study duration (up to 21 months)
Measure: Number; unit: BinaxNow Rapid Antigen COVID-19 Tests
Units Other Than Participants: BinaxNOW Rapid Antigen COVID-19 Tests
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Number analyzed (BinaxNOW Rapid Antigen COVID-19 Tests) | 3254
BinaxNow Rapid Antigen COVID-19 Tests
  Number of positive COVID-19 tests | 39
  Total number of tests performed | 3254

6. Primary Outcome: Change in False-positive Rate: Number of Negative Confirmatory Polymerase Chain Reaction (PCR) as Compared to Total PCR Run for COVID-19 Testing
Description: Data will be collected from parents via survey.
Time Frame: Study duration (up to 21 months)
Measure: Number; unit: Polymerase chain reaction for COVID-19
Units Other Than Participants: COVID-19 PCR Tests
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Number analyzed (COVID-19 PCR Tests) | 109
Polymerase chain reaction for COVID-19
  Number of negative confirmatory PCR tests | 1
  Total COVID-19 PCR tests | 109

7. Primary Outcome: Surveillance Opt in: Number of Participants Opting Into Surveillance Compared to Total Number of Enrolled Participants
Description: Data will be collected from parents via survey.
  - Caregivers were expected to test their child twice a week every week for the first three months. After that time, caregivers could opt-in to surveillance testing (expected testing twice a week every week) or proceed with symptomatic-only testing (no "expected" tests for caregivers).
Time Frame: At month 3
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Participants opting into surveillance testing | 32
  Participants not opting into surveillance testing | 19

8. Primary Outcome: Change in Susceptibility: Number of Fully Vaccinated People Who Interact With Participant's Child at School
Description: "How many of the people who interact with your child at school have been fully vaccinated?" Response options: "None", "A few", "Some" "Most", "All", "Don't Know" Dichotomized into: ("Most" or "All") vs. ("None", "A few", "Some", "Don't Know)
Time Frame: baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: "Most" or "All" of the people who interact with their child at school have been fully vaccinated | 12
  Baseline: "None", "A few", "Some", "Don't Know" | 39
  3-month: number analyzed (Participants) | 48
  3-month: "Most" or "All" of the people who interact with their child at school have been fully vaccinated | 9
  3-month: "None", "A few", "Some", "Don't Know" | 39
  6-month: number analyzed (Participants) | 46
  6-month: "Most" or "All" of the people who interact with their child at school have been fully vaccinated | 12
  6-month: "None", "A few", "Some", "Don't Know" | 34
  9-month: number analyzed (Participants) | 45
  9-month: "Most" or "All" of the people who interact with their child at school have been fully vaccinated | 10
  9-month: "None", "A few", "Some", "Don't Know" | 35
  15-month: number analyzed (Participants) | 39
  15-month: "Most" or "All" of the people who interact with their child at school have been fully vaccinated | 16
  15-month: "None", "A few", "Some", "Don't Know" | 23
  18-month: number analyzed (Participants) | 39
  18-month: "Most" or "All" of the people who interact with their child at school have been fully vaccinated | 15
  18-month: "None", "A few", "Some", "Don't Know" | 24
  21-month: number analyzed (Participants) | 41
  21-month: "Most" or "All" of the people who interact with their child at school have been fully vaccinated | 15
  21-month: "None", "A few", "Some", "Don't Know" | 26
  24-month: number analyzed (Participants) | 44
  24-month: "Most" or "All" of the people who interact with their child at school have been fully vaccinated | 17
  24-month: "None", "A few", "Some", "Don't Know" | 27

9. Primary Outcome: Change in Susceptibility: School Takes Precautions
Description: The following question from the Participant's perceived susceptibility survey will be answered dichotomously and presented qualitatively:
  * How comfortable are you with...the ability of your child's school to take all precautions to stop the spread of COVID-19?
  * Response options: "Not at all", "A little", "Somewhat", "Very", "Extremely"
  * Dichotomized into: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
Time Frame: baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: "Very" or "Extremely" comfortable | 24
  Baseline: "Not at all", "A little", or "Somewhat" comfortable | 27
  3 months: number analyzed (Participants) | 48
  3 months: "Very" or "Extremely" comfortable | 17
  3 months: "Not at all", "A little", or "Somewhat" comfortable | 31
  6 months: number analyzed (Participants) | 46
  6 months: "Very" or "Extremely" comfortable | 20
  6 months: "Not at all", "A little", or "Somewhat" comfortable | 26
  9-12 months: number analyzed (Participants) | 45
  9-12 months: "Very" or "Extremely" comfortable | 24
  9-12 months: "Not at all", "A little", or "Somewhat" comfortable | 21
  15 months: number analyzed (Participants) | 39
  15 months: "Very" or "Extremely" comfortable | 16
  15 months: "Not at all", "A little", or "Somewhat" comfortable | 23
  18 months: number analyzed (Participants) | 37
  18 months: "Very" or "Extremely" comfortable | 16
  18 months: "Not at all", "A little", or "Somewhat" comfortable | 21
  21 months: number analyzed (Participants) | 43
  21 months: "Very" or "Extremely" comfortable | 13
  21 months: "Not at all", "A little", or "Somewhat" comfortable | 30
  24 months: number analyzed (Participants) | 45
  24 months: "Very" or "Extremely" comfortable | 21
  24 months: "Not at all", "A little", or "Somewhat" comfortable | 24

10. Primary Outcome: Change in Susceptibility: Likely to Get COVID-19
Description: Following questions from the Participant's perceived susceptibility survey will be answered dichotomously (agree or disagree) and presented qualitatively.
  * In your opinion, how likely is your child to get sick with COVID-19 by attending school in-person?
  * Response options: "Not at all", "A little", "Somewhat", "Very", "Extremely"
  * Dichotomized into: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
Time Frame: baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: "Very" or "Extremely" likely | 22
  Baseline: "Not at all", "A little", or "Somewhat" likely | 29
  3 months: number analyzed (Participants) | 48
  3 months: "Very" or "Extremely" likely | 18
  3 months: "Not at all", "A little", or "Somewhat" likely | 30
  6 months: number analyzed (Participants) | 45
  6 months: "Very" or "Extremely" likely | 21
  6 months: "Not at all", "A little", or "Somewhat" likely | 24
  9 months: number analyzed (Participants) | 44
  9 months: "Very" or "Extremely" likely | 16
  9 months: "Not at all", "A little", or "Somewhat" likely | 28
  15 months: number analyzed (Participants) | 39
  15 months: "Very" or "Extremely" likely | 19
  15 months: "Not at all", "A little", or "Somewhat" likely | 20
  18 months: number analyzed (Participants) | 39
  18 months: "Very" or "Extremely" likely | 23
  18 months: "Not at all", "A little", or "Somewhat" likely | 16
  21 months: number analyzed (Participants) | 42
  21 months: "Very" or "Extremely" likely | 23
  21 months: "Not at all", "A little", or "Somewhat" likely | 19
  24 months: number analyzed (Participants) | 45
  24 months: "Very" or "Extremely" likely | 25
  24 months: "Not at all", "A little", or "Somewhat" likely | 20

11. Primary Outcome: Change in Percentage of Participants for Perceived Severity Survey Question: Health Severely Affected
Description: Parent survey perceived severity construct variables will include:
  * If your child was sick with COVID-19, how likely would...their health be severely affected
  * Response options: "Not at all", "A little", "Somewhat", "Very", "Extremely"
  * Dichotomized into: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
Time Frame: 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  15 month: number analyzed (Participants) | 38
  15 month: "Very" or "Extremely" likely | 20
  15 month: "Not at all", "A little", or "Somewhat" likely | 18
  18 month: number analyzed (Participants) | 39
  18 month: "Very" or "Extremely" likely | 25
  18 month: "Not at all", "A little", or "Somewhat" likely | 14
  21 month: number analyzed (Participants) | 43
  21 month: "Very" or "Extremely" likely | 29
  21 month: "Not at all", "A little", or "Somewhat" likely | 14
  24 month: number analyzed (Participants) | 45
  24 month: "Very" or "Extremely" likely | 26
  24 month: "Not at all", "A little", or "Somewhat" likely | 19

12. Primary Outcome: Change in Percentage of Participants to the Perceived Severity Survey Question: Health Permanently Reduced
Description: Parent survey perceived severity construct variables will be:
  * "If your child was sick with COVID-19, how likely would...their health be permanently reduced"
  * Response options: "Not at all", "A little", "Somewhat", "Very", "Extremely"
  * Dichotomized into: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
Time Frame: 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  15-month: number analyzed (Participants) | 38
  15-month: "Very" or "Extremely" likely | 17
  15-month: "Not at all", "A little", or "Somewhat" likely | 21
  18-month: number analyzed (Participants) | 39
  18-month: "Very" or "Extremely" likely | 20
  18-month: "Not at all", "A little", or "Somewhat" likely | 19
  21-month: number analyzed (Participants) | 43
  21-month: "Very" or "Extremely" likely | 18
  21-month: "Not at all", "A little", or "Somewhat" likely | 25
  24-month: number analyzed (Participants) | 45
  24-month: "Very" or "Extremely" likely | 19
  24-month: "Not at all", "A little", or "Somewhat" likely | 26

13. Primary Outcome: Change in Percentage of Participants to the Perceived Severity Survey Question: Grave Health Consequences
Description: Parent survey perceived severity construct variables will be:
  * "If my child was sick with COVID-19, they would have grave health consequences."
  * Response options: "Not at all", "A little", "Somewhat", "Very", "Extremely"
  * Dichotomized into: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
Time Frame: 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  15 month: number analyzed (Participants) | 38
  15 month: "Very" or "Extremely" likely | 17
  15 month: "Not at all", "A little", or "Somewhat" likely | 21
  18 month: number analyzed (Participants) | 39
  18 month: "Very" or "Extremely" likely | 21
  18 month: "Not at all", "A little", or "Somewhat" likely | 18
  21 month: number analyzed (Participants) | 43
  21 month: "Very" or "Extremely" likely | 19
  21 month: "Not at all", "A little", or "Somewhat" likely | 24
  24 month: number analyzed (Participants) | 44
  24 month: "Very" or "Extremely" likely | 20
  24 month: "Not at all", "A little", or "Somewhat" likely | 24

14. Primary Outcome: Change in Motivation to Attend School (Quite a Bit / A Great Deal vs. Not)
Description: Participants will answer the following survey question in quite a bit / a great deal vs not:
  * "Based on the situation right now, how much do you want your child to attend school in-person at least some of the time?"
Time Frame: Baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: "Quite a bit" or "A great deal" | 33
  Baseline: "Somewhat," "A little," or "Not at all" | 18
  3 month: number analyzed (Participants) | 48
  3 month: "Quite a bit" or "A great deal" | 29
  3 month: "Somewhat," "A little," or "Not at all" | 19
  6 month: number analyzed (Participants) | 46
  6 month: "Quite a bit" or "A great deal" | 29
  6 month: "Somewhat," "A little," or "Not at all" | 17
  9 month: number analyzed (Participants) | 45
  9 month: "Quite a bit" or "A great deal" | 35
  9 month: "Somewhat," "A little," or "Not at all" | 10
  15 month: number analyzed (Participants) | 39
  15 month: "Quite a bit" or "A great deal" | 28
  15 month: "Somewhat," "A little," or "Not at all" | 11
  18 month: number analyzed (Participants) | 39
  18 month: "Quite a bit" or "A great deal" | 27
  18 month: "Somewhat," "A little," or "Not at all" | 12
  21 month: number analyzed (Participants) | 42
  21 month: "Quite a bit" or "A great deal" | 33
  21 month: "Somewhat," "A little," or "Not at all" | 9
  24 month: number analyzed (Participants) | 45
  24 month: "Quite a bit" or "A great deal" | 35
  24 month: "Somewhat," "A little," or "Not at all" | 10

15. Primary Outcome: Change in Perceived Benefits to Attend School: Important to Health
Description: Parent survey perceived benefits construct survey will be having 6 questions ranging from benefits to child's overall health, therapy needs, impact on family. Survey will be analyzed qualitatively.
  * How important is attending school in-person to your child's overall health?
  * Dichotomized into: ("Not at all important", "A little important", "Somewhat important") vs. ("Very important", "Extremely important")
Time Frame: Baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: "Very important" or "Extremely important" | 37
  Baseline: "Not at all important", "A little important", or "Somewhat important" | 14
  3 month: number analyzed (Participants) | 48
  3 month: "Very important" or "Extremely important" | 29
  3 month: "Not at all important", "A little important", or "Somewhat important" | 19
  6 month: number analyzed (Participants) | 46
  6 month: "Very important" or "Extremely important" | 31
  6 month: "Not at all important", "A little important", or "Somewhat important" | 15
  9 month: number analyzed (Participants) | 45
  9 month: "Very important" or "Extremely important" | 34
  9 month: "Not at all important", "A little important", or "Somewhat important" | 11
  15 month: number analyzed (Participants) | 39
  15 month: "Very important" or "Extremely important" | 29
  15 month: "Not at all important", "A little important", or "Somewhat important" | 10
  18 month: number analyzed (Participants) | 39
  18 month: "Very important" or "Extremely important" | 31
  18 month: "Not at all important", "A little important", or "Somewhat important" | 8
  21 month: number analyzed (Participants) | 42
  21 month: "Very important" or "Extremely important" | 32
  21 month: "Not at all important", "A little important", or "Somewhat important" | 10
  24 month: number analyzed (Participants) | 44
  24 month: "Very important" or "Extremely important" | 29
  24 month: "Not at all important", "A little important", or "Somewhat important" | 15

16. Primary Outcome: Change in Perceived Benefits to Attend School: In-person Schooling
Description: Parent survey perceived benefits construct survey will be having 6 questions ranging from benefits to child's overall health, therapy needs, and impact on family. Survey will be analyzed qualitatively.
  * Compared to fully virtual school, how much better or worse is attending any school in-person for your child?
  * Dichotomized into: ("Quite a bit worse", "Somewhat worse", "A little bit worse", "Neither better nor worse") vs. ("A little bit better", "Somewhat better", "Quite a bit better")
Time Frame: Baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: number analyzed (Participants) | 50
  Baseline: "A little bit better", "Somewhat better", or "Quite a bit better" | 35
  Baseline: "Quite a bit worse", "Somewhat worse", "A little bit worse", or "Neither better nor worse" | 15
  3 month: number analyzed (Participants) | 48
  3 month: "A little bit better", "Somewhat better", or "Quite a bit better" | 33
  3 month: "Quite a bit worse", "Somewhat worse", "A little bit worse", or "Neither better nor worse" | 15
  6 month: number analyzed (Participants) | 46
  6 month: "A little bit better", "Somewhat better", or "Quite a bit better" | 32
  6 month: "Quite a bit worse", "Somewhat worse", "A little bit worse", or "Neither better nor worse" | 14
  9 month: number analyzed (Participants) | 45
  9 month: "A little bit better", "Somewhat better", or "Quite a bit better" | 35
  9 month: "Quite a bit worse", "Somewhat worse", "A little bit worse", or "Neither better nor worse" | 10
  15 month: number analyzed (Participants) | 39
  15 month: "A little bit better", "Somewhat better", or "Quite a bit better" | 32
  15 month: "Quite a bit worse", "Somewhat worse", "A little bit worse", or "Neither better nor worse" | 7
  18 month: number analyzed (Participants) | 39
  18 month: "A little bit better", "Somewhat better", or "Quite a bit better" | 29
  18 month: "Quite a bit worse", "Somewhat worse", "A little bit worse", or "Neither better nor worse" | 10
  21 month: number analyzed (Participants) | 43
  21 month: "A little bit better", "Somewhat better", or "Quite a bit better" | 37
  21 month: "Quite a bit worse", "Somewhat worse", "A little bit worse", or "Neither better nor worse" | 6
  24 month: number analyzed (Participants) | 45
  24 month: "A little bit better", "Somewhat better", or "Quite a bit better" | 36
  24 month: "Quite a bit worse", "Somewhat worse", "A little bit worse", or "Neither better nor worse" | 9

17. Primary Outcome: Change in Perceived Benefits to Attend School: Therapy Needs
Description: Parent survey perceived benefits construct survey will be having 6 questions ranging from benefits to child's overall health, therapy needs, impact on family. Survey will be analyzed qualitatively.
  * How much of your child's therapy needs are only met by attending school in-person?
  * Dichotomized into: ("None", "A few", "Some" vs. "Most", "All")
Time Frame: Baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: "Most", "All" | 38
  Baseline: "None", "A few", "Some" | 13
  3 month: number analyzed (Participants) | 48
  3 month: "Most", "All" | 32
  3 month: "None", "A few", "Some" | 16
  6 month: number analyzed (Participants) | 46
  6 month: "Most", "All" | 33
  6 month: "None", "A few", "Some" | 13
  9 month: number analyzed (Participants) | 45
  9 month: "Most", "All" | 31
  9 month: "None", "A few", "Some" | 14
  15 month: number analyzed (Participants) | 39
  15 month: "Most", "All" | 26
  15 month: "None", "A few", "Some" | 13
  18 month: number analyzed (Participants) | 39
  18 month: "Most", "All" | 27
  18 month: "None", "A few", "Some" | 12
  21 month: number analyzed (Participants) | 43
  21 month: "Most", "All" | 29
  21 month: "None", "A few", "Some" | 14
  24 month: number analyzed (Participants) | 45
  24 month: "Most", "All" | 30
  24 month: "None", "A few", "Some" | 15

18. Primary Outcome: Change in Perceived Benefits to Attend School: Positive for Family
Description: Parent survey perceived benefits construct survey will be having 6 questions ranging from benefits to child's overall health, therapy needs, impact on family. Survey will be analyzed qualitatively.
  * How positive or negative is your child attending school in-person for...your family
  * Dichotomized into: ("Very negative", "Somewhat negative", "A little negative", "Neutral") vs. ("A little positive", "Somewhat positive", "Very positive")
Time Frame: Baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: number analyzed (Participants) | 50
  Baseline: "A little positive", "Somewhat positive", or "Very positive" | 37
  Baseline: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 13
  3 month: number analyzed (Participants) | 48
  3 month: "A little positive", "Somewhat positive", or "Very positive" | 37
  3 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 11
  6 month: number analyzed (Participants) | 46
  6 month: "A little positive", "Somewhat positive", or "Very positive" | 38
  6 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 8
  9 month: number analyzed (Participants) | 45
  9 month: "A little positive", "Somewhat positive", or "Very positive" | 38
  9 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 7
  15 month: number analyzed (Participants) | 39
  15 month: "A little positive", "Somewhat positive", or "Very positive" | 31
  15 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 8
  18 month: number analyzed (Participants) | 39
  18 month: "A little positive", "Somewhat positive", or "Very positive" | 30
  18 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 9
  21 month: number analyzed (Participants) | 43
  21 month: "A little positive", "Somewhat positive", or "Very positive" | 36
  21 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 7
  24 month: number analyzed (Participants) | 45
  24 month: "A little positive", "Somewhat positive", or "Very positive" | 37
  24 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 8

19. Primary Outcome: Change in Perceived Benefits to Attend School: Positive for Staff
Description: Parent survey perceived benefits construct survey will be having 6 questions ranging from benefits to child's overall health, therapy needs, impact on family. Survey will be analyzed qualitatively.
  * How positive or negative is your child attending school in-person for...the staff and teachers
  * Dichotomized into: ("Very negative", "Somewhat negative", "A little negative", "Neutral") vs. ("A little positive", "Somewhat positive", "Very positive")
Time Frame: Baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: number analyzed (Participants) | 50
  Baseline: "A little positive", "Somewhat positive", or "Very positive" | 34
  Baseline: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 16
  3 month: number analyzed (Participants) | 47
  3 month: "A little positive", "Somewhat positive", or "Very positive" | 36
  3 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 11
  6 month: number analyzed (Participants) | 46
  6 month: "A little positive", "Somewhat positive", or "Very positive" | 32
  6 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 14
  9 month: number analyzed (Participants) | 45
  9 month: "A little positive", "Somewhat positive", or "Very positive" | 38
  9 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 7
  15 month: number analyzed (Participants) | 39
  15 month: "A little positive", "Somewhat positive", or "Very positive" | 28
  15 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 11
  18 month: number analyzed (Participants) | 39
  18 month: "A little positive", "Somewhat positive", or "Very positive" | 30
  18 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 9
  21 month: number analyzed (Participants) | 43
  21 month: "A little positive", "Somewhat positive", or "Very positive" | 36
  21 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 7
  24 month: number analyzed (Participants) | 45
  24 month: "A little positive", "Somewhat positive", or "Very positive" | 36
  24 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 9

20. Primary Outcome: Change in Perceived Benefits to Attend School: Keep Jobs
Description: Parent survey perceived benefits construct survey will be having 6 questions ranging from benefits to child's overall health, therapy needs, impact on family. Survey will be analyzed qualitatively.
  * Does your child attending school in-person help the adults in your family to keep their jobs?
  * Response options: Yes / No
Time Frame: Baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: Yes | 32
  Baseline: No | 19
  3 month: number analyzed (Participants) | 48
  3 month: Yes | 29
  3 month: No | 19
  6 month: number analyzed (Participants) | 46
  6 month: Yes | 26
  6 month: No | 20
  9 month: number analyzed (Participants) | 45
  9 month: Yes | 24
  9 month: No | 21
  15 month: number analyzed (Participants) | 39
  15 month: Yes | 22
  15 month: No | 17
  18 month: number analyzed (Participants) | 39
  18 month: Yes | 25
  18 month: No | 14
  21 month: number analyzed (Participants) | 43
  21 month: Yes | 29
  21 month: No | 14
  24 month: number analyzed (Participants) | 45
  24 month: Yes | 28
  24 month: No | 17

21. Primary Outcome: Change in Barriers to School Attendance: Number of People
Description: Survey will have following questions which will be answered dichotomously very/extremely [comfortable] vs not.
  * How comfortable are you with the number of people around your child at school?
  * Dichotomized into: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
Time Frame: baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: "Very" or "Extremely" comfortable | 21
  Baseline: "Not at all", "A little", or "Somewhat" comfortable | 30
  3 month: number analyzed (Participants) | 48
  3 month: "Very" or "Extremely" comfortable | 14
  3 month: "Not at all", "A little", or "Somewhat" comfortable | 34
  6 month: number analyzed (Participants) | 46
  6 month: "Very" or "Extremely" comfortable | 17
  6 month: "Not at all", "A little", or "Somewhat" comfortable | 29
  9 month: number analyzed (Participants) | 45
  9 month: "Very" or "Extremely" comfortable | 19
  9 month: "Not at all", "A little", or "Somewhat" comfortable | 26
  15 month: number analyzed (Participants) | 39
  15 month: "Very" or "Extremely" comfortable | 12
  15 month: "Not at all", "A little", or "Somewhat" comfortable | 27
  18 month: number analyzed (Participants) | 39
  18 month: "Very" or "Extremely" comfortable | 14
  18 month: "Not at all", "A little", or "Somewhat" comfortable | 25
  21 month: number analyzed (Participants) | 43
  21 month: "Very" or "Extremely" comfortable | 13
  21 month: "Not at all", "A little", or "Somewhat" comfortable | 30
  24 month: number analyzed (Participants) | 45
  24 month: "Very" or "Extremely" comfortable | 15
  24 month: "Not at all", "A little", or "Somewhat" comfortable | 30

22. Primary Outcome: Change in Barriers to School Attendance: Proximity
Description: Survey will have following questions which will be answered dichotomously very/extremely [comfortable] vs not.
  * How comfortable are you with how close people have to be to your child at school?
  * Dichotomized into: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
Time Frame: Baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: number analyzed (Participants) | 50
  Baseline: "Very" or "Extremely" comfortable | 18
  Baseline: "Not at all", "A little", or "Somewhat" comfortable | 32
  3 month: number analyzed (Participants) | 48
  3 month: "Very" or "Extremely" comfortable | 12
  3 month: "Not at all", "A little", or "Somewhat" comfortable | 36
  6 month: number analyzed (Participants) | 46
  6 month: "Very" or "Extremely" comfortable | 18
  6 month: "Not at all", "A little", or "Somewhat" comfortable | 28
  9 month: number analyzed (Participants) | 45
  9 month: "Very" or "Extremely" comfortable | 17
  9 month: "Not at all", "A little", or "Somewhat" comfortable | 28
  15 month: number analyzed (Participants) | 39
  15 month: "Very" or "Extremely" comfortable | 11
  15 month: "Not at all", "A little", or "Somewhat" comfortable | 28
  18 month: number analyzed (Participants) | 39
  18 month: "Very" or "Extremely" comfortable | 13
  18 month: "Not at all", "A little", or "Somewhat" comfortable | 26
  21 month: number analyzed (Participants) | 43
  21 month: "Very" or "Extremely" comfortable | 12
  21 month: "Not at all", "A little", or "Somewhat" comfortable | 31
  24 month: number analyzed (Participants) | 45
  24 month: "Very" or "Extremely" comfortable | 18
  24 month: "Not at all", "A little", or "Somewhat" comfortable | 27

23. Primary Outcome: Change in Barriers to School Attendance: PPE
Description: Survey will have following questions which will be answered dichotomously very/extremely [comfortable] vs not.
  * How comfortable are you with the amount personal protective equipment (PPE), such as masks and gloves, available at school?
  * Dichotomized into: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
Time Frame: Baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: "Very" or "Extremely" comfortable | 24
  Baseline: "Not at all", "A little", or "Somewhat" comfortable | 27
  3 month: number analyzed (Participants) | 48
  3 month: "Very" or "Extremely" comfortable | 20
  3 month: "Not at all", "A little", or "Somewhat" comfortable | 28
  6 month: number analyzed (Participants) | 46
  6 month: "Very" or "Extremely" comfortable | 25
  6 month: "Not at all", "A little", or "Somewhat" comfortable | 21
  9 month: number analyzed (Participants) | 45
  9 month: "Very" or "Extremely" comfortable | 20
  9 month: "Not at all", "A little", or "Somewhat" comfortable | 25
  15 month: number analyzed (Participants) | 39
  15 month: "Very" or "Extremely" comfortable | 10
  15 month: "Not at all", "A little", or "Somewhat" comfortable | 29
  18 month: number analyzed (Participants) | 39
  18 month: "Very" or "Extremely" comfortable | 21
  18 month: "Not at all", "A little", or "Somewhat" comfortable | 18
  21 month: number analyzed (Participants) | 43
  21 month: "Very" or "Extremely" comfortable | 19
  21 month: "Not at all", "A little", or "Somewhat" comfortable | 24
  24 month: number analyzed (Participants) | 45
  24 month: "Very" or "Extremely" comfortable | 21
  24 month: "Not at all", "A little", or "Somewhat" comfortable | 24

24. Primary Outcome: Change in Barriers to School Attendance: Testing
Description: Survey will have following questions which will be answered dichotomously very/extremely [comfortable] vs not.
  * How comfortable are you with the amount of COVID-19 testing among school staff and classmates?
  * Dichotomized into: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
Time Frame: Baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: "Very" or "Extremely" comfortable | 11
  Baseline: "Not at all", "A little", or "Somewhat" comfortable | 40
  3 month: number analyzed (Participants) | 48
  3 month: "Very" or "Extremely" comfortable | 14
  3 month: "Not at all", "A little", or "Somewhat" comfortable | 34
  6 month: number analyzed (Participants) | 45
  6 month: "Very" or "Extremely" comfortable | 16
  6 month: "Not at all", "A little", or "Somewhat" comfortable | 29
  9 month: number analyzed (Participants) | 44
  9 month: "Very" or "Extremely" comfortable | 18
  9 month: "Not at all", "A little", or "Somewhat" comfortable | 26
  15 month: number analyzed (Participants) | 39
  15 month: "Very" or "Extremely" comfortable | 10
  15 month: "Not at all", "A little", or "Somewhat" comfortable | 29
  18 month: number analyzed (Participants) | 39
  18 month: "Very" or "Extremely" comfortable | 13
  18 month: "Not at all", "A little", or "Somewhat" comfortable | 26
  21 month: number analyzed (Participants) | 43
  21 month: "Very" or "Extremely" comfortable | 13
  21 month: "Not at all", "A little", or "Somewhat" comfortable | 30
  24 month: number analyzed (Participants) | 45
  24 month: "Very" or "Extremely" comfortable | 15
  24 month: "Not at all", "A little", or "Somewhat" comfortable | 30

25. Primary Outcome: Change in Barriers to School Attendance: Following Recommendations
Description: Survey will have following questions which will be answered dichotomously very/extremely [comfortable] vs not.
  * How comfortable are you with how closely parents of classmates follow recommendations to keep your child safe?
  * Dichotomized into: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
Time Frame: Baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: "Very" or "Extremely" comfortable | 13
  Baseline: "Not at all", "A little", or "Somewhat" comfortable | 38
  3 month: number analyzed (Participants) | 48
  3 month: "Very" or "Extremely" comfortable | 15
  3 month: "Not at all", "A little", or "Somewhat" comfortable | 33
  6 month: number analyzed (Participants) | 46
  6 month: "Very" or "Extremely" comfortable | 14
  6 month: "Not at all", "A little", or "Somewhat" comfortable | 32
  9 month: number analyzed (Participants) | 45
  9 month: "Very" or "Extremely" comfortable | 14
  9 month: "Not at all", "A little", or "Somewhat" comfortable | 31
  15 month: number analyzed (Participants) | 39
  15 month: "Very" or "Extremely" comfortable | 9
  15 month: "Not at all", "A little", or "Somewhat" comfortable | 30
  18 month: number analyzed (Participants) | 39
  18 month: "Very" or "Extremely" comfortable | 13
  18 month: "Not at all", "A little", or "Somewhat" comfortable | 26
  21 month: number analyzed (Participants) | 43
  21 month: "Very" or "Extremely" comfortable | 11
  21 month: "Not at all", "A little", or "Somewhat" comfortable | 32
  24 month: number analyzed (Participants) | 45
  24 month: "Very" or "Extremely" comfortable | 14
  24 month: "Not at all", "A little", or "Somewhat" comfortable | 31

26. Primary Outcome: Change in Barriers to School Attendance: Transportation
Description: Survey will have following questions which will be answered dichotomously very/extremely vs not.
  * How difficult is it to transport your child to or from school as a result of COVID-19?
  * Dichotomized as: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
Time Frame: Baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: "Very" or "Extremely" difficult | 5
  Baseline: "Not at all", "A little", or "Somewhat" difficult | 46
  3 month: number analyzed (Participants) | 48
  3 month: "Very" or "Extremely" difficult | 1
  3 month: "Not at all", "A little", or "Somewhat" difficult | 47
  6 month: number analyzed (Participants) | 46
  6 month: "Very" or "Extremely" difficult | 3
  6 month: "Not at all", "A little", or "Somewhat" difficult | 43
  9 month: number analyzed (Participants) | 45
  9 month: "Very" or "Extremely" difficult | 4
  9 month: "Not at all", "A little", or "Somewhat" difficult | 41
  15 month: number analyzed (Participants) | 39
  15 month: "Very" or "Extremely" difficult | 4
  15 month: "Not at all", "A little", or "Somewhat" difficult | 35
  18 month: number analyzed (Participants) | 37
  18 month: "Very" or "Extremely" difficult | 2
  18 month: "Not at all", "A little", or "Somewhat" difficult | 35
  21 month: number analyzed (Participants) | 43
  21 month: "Very" or "Extremely" difficult | 2
  21 month: "Not at all", "A little", or "Somewhat" difficult | 41
  24 month: number analyzed (Participants) | 45
  24 month: "Very" or "Extremely" difficult | 1
  24 month: "Not at all", "A little", or "Somewhat" difficult | 44

27. Primary Outcome: Change in Barriers to School Attendance: Wash
Description: Survey will have following questions which will be answered dichotomously very/extremely vs not.
  * In your child's school, do they have access to necessary facilities to wash?
  * Dichotomized as: ("Yes, all of the time", "Yes, most of the time") vs. ("Some of the time", "Rarely", "Not at all")
Time Frame: Baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: "Yes, all of the time" or "Yes, most of the time" | 43
  Baseline: "Some of the time", "Rarely", or "Not at all" | 8
  3 month: number analyzed (Participants) | 48
  3 month: "Yes, all of the time" or "Yes, most of the time" | 45
  3 month: "Some of the time", "Rarely", or "Not at all" | 3
  6 month: number analyzed (Participants) | 46
  6 month: "Yes, all of the time" or "Yes, most of the time" | 41
  6 month: "Some of the time", "Rarely", or "Not at all" | 5
  9 month: number analyzed (Participants) | 45
  9 month: "Yes, all of the time" or "Yes, most of the time" | 40
  9 month: "Some of the time", "Rarely", or "Not at all" | 5
  15 month: number analyzed (Participants) | 39
  15 month: "Yes, all of the time" or "Yes, most of the time" | 33
  15 month: "Some of the time", "Rarely", or "Not at all" | 6
  18 month: number analyzed (Participants) | 39
  18 month: "Yes, all of the time" or "Yes, most of the time" | 32
  18 month: "Some of the time", "Rarely", or "Not at all" | 7
  21 month: number analyzed (Participants) | 43
  21 month: "Yes, all of the time" or "Yes, most of the time" | 37
  21 month: "Some of the time", "Rarely", or "Not at all" | 6
  24 month: number analyzed (Participants) | 45
  24 month: "Yes, all of the time" or "Yes, most of the time" | 39
  24 month: "Some of the time", "Rarely", or "Not at all" | 6

28. Primary Outcome: Change in Barriers to School Attendance: Close Contact
Description: Survey will have following questions which will be answered dichotomously very/extremely [comfortable] vs not.
  * While in school, is your child required to be in close contact (i.e., within 6 ft) with others? 'Others' includes teachers, aides, nurses, and classmates.
  * Dichotomized as: ("Yes, all of the time", "Yes, most of the time") vs. ("Some of the time", "Rarely", "Not at all")
Time Frame: Baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: "Yes, all of the time" or "Yes, most of the time" | 47
  Baseline: "Some of the time", "Rarely", or "Not at all" | 4
  3 month: number analyzed (Participants) | 48
  3 month: "Yes, all of the time" or "Yes, most of the time" | 42
  3 month: "Some of the time", "Rarely", or "Not at all" | 6
  6 month: number analyzed (Participants) | 46
  6 month: "Yes, all of the time" or "Yes, most of the time" | 41
  6 month: "Some of the time", "Rarely", or "Not at all" | 5
  9 month: number analyzed (Participants) | 45
  9 month: "Yes, all of the time" or "Yes, most of the time" | 44
  9 month: "Some of the time", "Rarely", or "Not at all" | 1
  15 month: number analyzed (Participants) | 39
  15 month: "Yes, all of the time" or "Yes, most of the time" | 36
  15 month: "Some of the time", "Rarely", or "Not at all" | 3
  18 month: number analyzed (Participants) | 39
  18 month: "Yes, all of the time" or "Yes, most of the time" | 36
  18 month: "Some of the time", "Rarely", or "Not at all" | 3
  21 month: number analyzed (Participants) | 43
  21 month: "Yes, all of the time" or "Yes, most of the time" | 40
  21 month: "Some of the time", "Rarely", or "Not at all" | 3
  24 month: number analyzed (Participants) | 44
  24 month: "Yes, all of the time" or "Yes, most of the time" | 43
  24 month: "Some of the time", "Rarely", or "Not at all" | 1

29. Primary Outcome: Change in Barriers to School Attendance: Masking
Description: Survey will have following questions which will be answered dichotomously very/extremely vs not.
  * While in school, is your child able to wear a mask?
  * Dichotomized as: ("Yes, all of the time", "Yes, most of the time") vs. ("Some of the time", "Rarely", "Not at all")
Time Frame: Baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: "Yes, all of the time" or "Yes, most of the time" | 24
  Baseline: "Some of the time", "Rarely", or "Not at all" | 27
  3 month: number analyzed (Participants) | 48
  3 month: "Yes, all of the time" or "Yes, most of the time" | 23
  3 month: "Some of the time", "Rarely", or "Not at all" | 25
  6 month: number analyzed (Participants) | 46
  6 month: "Yes, all of the time" or "Yes, most of the time" | 21
  6 month: "Some of the time", "Rarely", or "Not at all" | 25
  9 month: number analyzed (Participants) | 45
  9 month: "Yes, all of the time" or "Yes, most of the time" | 19
  9 month: "Some of the time", "Rarely", or "Not at all" | 26
  15 month: number analyzed (Participants) | 39
  15 month: "Yes, all of the time" or "Yes, most of the time" | 18
  15 month: "Some of the time", "Rarely", or "Not at all" | 21
  18 month: number analyzed (Participants) | 39
  18 month: "Yes, all of the time" or "Yes, most of the time" | 16
  18 month: "Some of the time", "Rarely", or "Not at all" | 23
  21 month: number analyzed (Participants) | 43
  21 month: "Yes, all of the time" or "Yes, most of the time" | 14
  21 month: "Some of the time", "Rarely", or "Not at all" | 29
  24 month: number analyzed (Participants) | 44
  24 month: "Yes, all of the time" or "Yes, most of the time" | 16
  24 month: "Some of the time", "Rarely", or "Not at all" | 28

30. Primary Outcome: Change in Cues: Has a Teacher or Staff Member Encouraged Child to Attend School In-person? (Y/N)
Description: Participants will answer the following survey question in Yes/No:
  * "Teachers/staff have asked for my child to attend school."- Y/N
Time Frame: baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: Yes | 29
  Baseline: No | 22
  3-month: number analyzed (Participants) | 48
  3-month: Yes | 31
  3-month: No | 17
  6-month: number analyzed (Participants) | 46
  6-month: Yes | 34
  6-month: No | 12
  9-month: number analyzed (Participants) | 45
  9-month: Yes | 32
  9-month: No | 13
  15-month: number analyzed (Participants) | 39
  15-month: Yes | 25
  15-month: No | 14
  18-month: number analyzed (Participants) | 39
  18-month: Yes | 30
  18-month: No | 9
  21-month: number analyzed (Participants) | 43
  21-month: Yes | 33
  21-month: No | 10
  24-month: number analyzed (Participants) | 44
  24-month: Yes | 36
  24-month: No | 8

31. Primary Outcome: Change in Option and Practice: Currently, is Child Attending School In-person, Either Full-time or as Part of a Hybrid or Part-time Schedule? Y/N
Description: Participant will be asked the attendance question in survey. It will be answered in Yes/No
Time Frame: baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: Yes | 29
  Baseline: No | 22
  3-month: number analyzed (Participants) | 48
  3-month: Yes | 35
  3-month: No | 13
  6-month: number analyzed (Participants) | 46
  6-month: Yes | 35
  6-month: No | 11
  9-month: number analyzed (Participants) | 45
  9-month: Yes | 37
  9-month: No | 8
  15-month: number analyzed (Participants) | 39
  15-month: Yes | 32
  15-month: No | 7
  18-month: number analyzed (Participants) | 39
  18-month: Yes | 33
  18-month: No | 6
  21-month: number analyzed (Participants) | 43
  21-month: Yes | 37
  21-month: No | 6
  24-month: number analyzed (Participants) | 45
  24-month: Yes | 38
  24-month: No | 7

32. Primary Outcome: Change in Option and Practice: Currently, if Participant Wanted, Could the Child Attend School In-person, Either Full-time or as Part of a Hybrid or Part-time Schedule? Y/N
Description: Participant will be asked the attendance question in survey. It will be answered in Yes/No.
  Survey branching logic asked this question only to participants whose child was not currently attending school in person, either full-time or as part of a hybrid or part-time schedule. The number analyzed represents the number of participants that answered this question.
Time Frame: baseline, 3 month, 6 month, 9-12 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver of Children With Medical Complexity (CMC)
Number analyzed (Participants) | 51
Participants
  Baseline: number analyzed (Participants) | 22
  Baseline: Yes | 14
  Baseline: No | 8
  3-month: number analyzed (Participants) | 13
  3-month: Yes | 9
  3-month: No | 4
  6-month: number analyzed (Participants) | 11
  6-month: Yes | 8
  6-month: No | 3
  9-month: number analyzed (Participants) | 8
  9-month: Yes | 7
  9-month: No | 1
  15-month: number analyzed (Participants) | 7
  15-month: Yes | 4
  15-month: No | 3
  18-month: number analyzed (Participants) | 6
  18-month: Yes | 3
  18-month: No | 3
  21-month: number analyzed (Participants) | 6
  21-month: Yes | 4
  21-month: No | 2
  24-month: number analyzed (Participants) | 7
  24-month: Yes | 4
  24-month: No | 3

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during active study participation, from enrollment to study exit, an average of 2 years, (study time frame = 4/2021 to 6/2023); any reportable events are followed to completion. Only children were assessed for AEs. Caregivers were not followed for AEs.
Description: Per protocol, any information disclosed to or discovered by staff indicating an undesirable experience associated with study participation will be reported to PI ASAP. PI determines if it's associated with study medical product and/or study procedures. Associated events will be reported to the IRB per local guidelines: https://irb.wisc.edu/wp-content/uploads/sites/2/sites/2/2022/07/AEdecisionguidewithFDAVAupdate_10_31_17.pdf. Additionally, events are documented in study files as Note-to-File.
Groups:
- Children With Medical Complexity (CMC): BinaxNOW Rapid Antigen System: BinaxNOW Rapid Antigen System (Abbott) is a point-of-care, lateral flow immunoassay intended for the qualitative detection of nucleocapsid protein antigen from SARS-CoV-2 in direct anterior nasal (nares) swabs. Internal controls are built into the testing system and results are available in 15 minutes.
  The use of the BinaxNOW system is authorized under the Food and Drug Administration's Emergency Use Authorization. The test is allowed for over-the-counter, non-prescription use with or without symptoms. The test may be used with children two years and older with the help of sample collection by an adult, and the test may be self-administered by anyone aged 15 years or more.
Arm/Group | Children With Medical Complexity (CMC)
All-Cause Mortality (participants affected / at risk) | 1/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT04895085/Prot_SAP_002.pdf
  • Informed Consent Form (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT04895085/ICF_000.pdf